CLINICAL TRIAL: NCT03109561
Title: APOE, Metabolism and Cognitive Function: An Assessment Via Indirect Calorimetry
Brief Title: Apolipoprotein E (ApoE) and Metabolism
Status: Completed | Type: Observational
Sponsor: Lance Johnson (Other)
Responsible Party: Sponsor-Investigator, Lance Johnson, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 17-0202-F1G
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Cognitive Function; Healthy
MeSH Terms: interventions — Apolipoproteins E; Metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 tablespoons of blood for DNA Testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Resting State Indirect Calorimetry — The investigator will measure the amount of oxygen participants breathe in and the amount of carbon dioxide they breathe out using a portable unit. Participants will be asked wearing a loose-fitting face mask that measures oxygen intake and carbon dioxide output.
Genetic: ApoE — The investigator will conduct a genetic test on DNA isolated from from the participants blood. Participants will be asked to provide about 2 tablespoons.
Diagnostic Test: Metabolism — To more accurately measure the amount of carbohydrates, fats and proteins that the participants bodies metabolize, participants will be asked to provide two urine samples (one at the beginning, and one at the end, of the study). The total amount of urine to be collected is approximately 4 teaspoons.
Other: Cognitive Challenge — Participants will be asked to follow simple instructions that are displayed on computer screen.

SUMMARY:
Impaired metabolism and the gene apolipoprotein E (ApoE) are independent risk factors for cognitive impairment and dementia. In humans, there are three major versions of apoE (E): E2, E3, and E4. Some studies suggest that the different versions of apoE have varying effects on whole body and brain metabolism. The goal of this project is to better understand the relationship between apoE and metabolism. This will help investigators identify new targets for the prevention and treatment of cognitive decline and dementia.

DETAILED DESCRIPTION:
The investigator hopes determine whether a participant's version of ApoE affects their metabolic rate at rest and during a cognitive challenge. To determine this, the investigator will measure basal (resting) metabolic rates using a technique called indirect calorimetry (IC). This is accomplished by wearing a loose-fitting face mask that measures oxygen intake and carbon dioxide output.

To more accurately measure the amount of carbohydrates, fats and proteins that the body is metabolizing, participants will be asked to provide two urine samples (one at the beginning, and one at the end, of the study).

To determine what version of ApoE the participant inherited, the investigator will conduct a genetic test on DNA isolated from the participant's blood.

ELIGIBILITY:
Inclusion Criteria:

* all races/ethnicities
* ages 18-65
* cognitively normal
* good health

Exclusion Criteria:

* pregnant or breastfeeding.
* have a bleeding disorder,
* have a history of stroke, seizures, Parkinson's disease, history of head injury with loss of consciousness, or other dementing disorder.
* have a history of alcoholism or drug abuse
* have a history of schizophrenia or currently suffer from bipolar disorder or major depression.
* have vision or hearing loss severe enough to interfere with cognitive testing

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cognitively normal and are in good overall health.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Indirect Calorimetry | 4 hours
  Measure resting state respiratory quotient in cognitively normal participants with various ApoE genotypes

SECONDARY OUTCOMES:
Respiratory Quotient (RQ) | 4 hours
  Measure RQ during a cognitive challenge in cognitively normal individuals with various ApoE genotypes

OTHER OUTCOMES:
Urea Nitrogen Output | 4 hours
  Improve RQ measure accuracy by determining urinary urea nitrogen output in collected urine samples from these subjects.
Genotype | 4 hours
  Genotype subjects using DNA isolated from collected blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Johnson1, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No